CLINICAL TRIAL: NCT00019552
Title: A Phase II Study of MGI-114 in Patients With Recurrent or Persistent Epithelial Ovarian Cancer
Brief Title: Irofulven in Treating Patients With Recurrent or Persistent Ovarian, Fallopian Tube, or Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066696; NCI-98-C-0162; MB-403; NCI-T98-0030
Record Dates: First submitted 2001-07-11; First posted 2004-04-13 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2002-01

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — irofulven

INTERVENTIONS:
Drug: irofulven

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of irofulven in treating patients who have recurrent or persistent ovarian, fallopian tube, or peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the clinical activity of irofulven in patients with recurrent or persistent ovarian epithelial cancer. II. Characterize the pharmacokinetic profile of this drug in these patients. III. Determine the pharmacodynamic relationship between plasma concentrations and clinical activity or toxicity of this drug in these patients.

OUTLINE: Patients are stratified according to the number of prior treatment regimens (1-2 vs 3 or more). Patients receive irofulven IV over 5 minutes on days 1-5. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients are followed every 4 weeks until death.

PROJECTED ACCRUAL: A maximum of 74 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent or persistent ovarian epithelial cancer, primary fallopian tube cancer, or primary peritoneal cancer that failed prior standard chemotherapy Measurable disease No history of brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Greater than 2 months Hematopoietic: Granulocyte count at least 1,500/mm3 Hemoglobin at least 9.0 g/dL (transfusion allowed) Platelet count at least 100,000/mm3 Hepatic: Bilirubin normal ALT and AST no greater than 2.5 times normal PT or PTT no greater than 1.5 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 50 mL/min Urinalysis normal BUN normal Electrolytes normal Cardiovascular: No unstable or newly diagnosed angina pectoris within the past 6 months No myocardial infarction within the past 6 months No New York Heart Association class II-IV congestive heart failure Pulmonary: No chronic obstructive lung disease requiring oxygen supplementation therapy or medication Other: No medical or surgical complications requiring intervention, such as: Impending bowel obstruction Active infection No other life-threatening illness No non-skin malignancy or melanoma within the past 4.5 years except curatively treated other malignancy with low risk of recurrence or surgically cured stage I endometrial cancer No uncontrolled seizures Not pregnant or nursing HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: Recovered from prior biologic therapy No prior bone marrow transplantation Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) Endocrine therapy: Recovered from prior endocrine therapy Radiotherapy: Recovered from prior radiotherapy No prior external beam radiotherapy Surgery: Recovered from prior surgery Other: At least 1 week since prior antibiotics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-09; Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gisele A. Sarosy, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Medicine Branch, Bethesda, Maryland, United States